CLINICAL TRIAL: NCT01561651
Title: Left Atrial Appendage Occlusion Study III
Acronym: LAAOS III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Principal Investigator, Richard Whitlock, Assistant Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LAAOSIII-2012
Record Dates: First submitted 2012-03-20; First posted 2012-03-23 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Cardiac Surgery With Cardiopulmonary Bypass; Atrial Fibrillation
Keywords: cardiac surgery; left atrial appendage; atrial fibrillation; stroke; non-CNS systemic embolism
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Left Atrial Appendage Occlusion Group (Experimental): Surgeon will close the left atrial appendage using a suture and/or a surgical stapler or a regulatory approved atrial appendage closure device during the patient's cardiac surgery procedure.
  Interventions: Other: Left Atrial Appendage Occlusion
- No Left Atrial Appendage Occlusion Group (No Intervention): Surgeon will not close the left atrial appendage during the patient's cardiac surgery procedure. Patient will be treated as per best medical practice for stroke prevention in atrial fibrillation. Treatment will be decided by the patient's primary care physician.

INTERVENTIONS:
Other: Left Atrial Appendage Occlusion — Surgeon will occlude the left atrial appendage using a suture and/or a surgical stapler or a regulatory approved atrial appendage closure during the patient's cardiac surgery procedure.
  Arms: Left Atrial Appendage Occlusion Group

SUMMARY:
Atrial fibrillation (AF) is a common heart rhythm disorder that leads to one-sixth of all strokes. Prevention of strokes in AF is achieved through the use of blood thinners such as coumadin. Although these blood thinners are effective, they are limited by the risk of serious bleeding, by physician and patient reluctance to use, and by noncompliance and discontinuation. The left atrial appendage is a structure on the upper chamber of the heart that is the most common source of stroke in patients with AF. This structure is easily accessible during open heart surgery for removal, and has been an area of interest for stroke prevention. However, there is currently no strong evidence that removing it works.

The LAAOS III trial will randomly (like the flip of a coin) assign patients with AF undergoing heart surgery for other reasons to have the left atrial appendage removed or not. These patients, other than this small procedure which has been shown to be quite safe, will be treated in the usual manner. The full study of 4700 patients, followed for an average of 4 years, will determine if removing the left atrial appendage can reduce stroke and other complications on top of usual therapy. A positive study will change the way heart surgery is performed on AF patients and results in a large reduction in the number of strokes in a large population. Further, it will promote further research into this approach that could be applied beyond AF patients undergoing heart surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 18 years of age
2. Undergoing a clinically indicated cardiac surgical procedure with the use of cardiopulmonary bypass
3. Have a documented history of atrial fibrillation or atrial flutter
4. CHA2DS2-VASc score ≥ 2
5. Have provided informed consent

Exclusion Criteria:

1. Patients undergoing off-pump cardiac surgery
2. Patients undergoing any of the following procedures:

   * heart transplant
   * complex congenital heart surgery
   * sole indication for surgery is ventricular assist device insertion
   * previous cardiac surgery requiring opening of the pericardium
   * mechanical valve implant
3. Patients who have had a previous placement of a percutaneous left atrial appendage closure device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4812 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Stroke or systemic arterial embolism | Common termination point (median follow-up of 4 years)
  First occurrence of ischemic stroke or transient ischemic attack with positive neuroimaging or systemic arterial embolism

SECONDARY OUTCOMES:
All cause stroke or transient ischemic attack with positive neuroimaging or systemic arterial embolism | Common termination point (median follow-up of 4 years)
  All cause stroke or transient ischemic attack with positive neuroimaging or systemic arterial embolism
Ischemic stroke or transient ischemic attack with positive neuroimaging or systemic arterial embolism or death | Common termination point (median follow-up of 4 years)
  Ischemic stroke* or transient ischemic attack with positive neuroimaging or systemic arterial embolism or death
Ischemic stroke or transient ischemic attack with positive neuroimaging or systemic arterial embolism > 30 days after surgery | Common termination point (median follow-up of 4 years)
  Ischemic stroke or transient ischemic attack with positive neuroimaging or systemic arterial embolism > 30 days after surgery
Total mortality | Common termination point (median follow-up of 4 years)
  Total mortality

OTHER OUTCOMES:
Readmission for heart failure | Common termination point (median follow-up of 4 years)
  Readmission for heart failure
Post-operative safety outcomes | 30 days post-surgery
  Operative safety outcomes (30-day mortality, chest tube output in the first post-operative 24 hours, rate of post-operative re-exploration for bleeding)
Major bleeding | Common termination point (median follow-up of 4 years)
  Major bleeding
Myocardial infarction | Common termination point (median follow-up of 4 years)
  Myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Richard Whitlock, MD, Principal Investigator — Population Health Research Institute/McMaster University; Stuart Connolly, MD, PhD, Study Chair — Population Health Research Institute/McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Katsanos AH, Whitlock RP, Belley-Cote EP, Brady K, Wang A, Srivastava A, Jacquin G, Weiss V, Volny O, Sramek M, Peeters A, Marto JP, Wrona P, Tsolaki A, Li L, Nucera A, Mikulik R, Perera K, Catanese L, Shoamanesh A, Sharma M. Stroke Mechanism and Severity After Left Atrial Appendage Occlusion: Insights From the LAAOS III Randomized Clinical Trial. JAMA Neurol. 2026 Jan 1;83(1):76-82. doi: 10.1001/jamaneurol.2025.4478. PMID 41247709
- [Derived] Kim KS, Belley-Cote EP, Walsh M, Wang A, Balasubramanian K, Treleaven N, Garg AX, Guyatt G, Whitlock RP. Left atrial appendage occlusion study III-Kidney substudy. Am Heart J. 2025 Oct;288:90-100. doi: 10.1016/j.ahj.2025.04.018. Epub 2025 Apr 19. PMID 40258408
- [Derived] Krisai P, Belley-Cote EP, McIntyre WF, Wong J, Tsiplova K, Brady K, Joseph P, Johansson I, Johnson L, Xing LY, Colli A, McGuinness S, Punjabi P, Reents W, Rega F, Budera P, Royse AG, Paparella D, Connolly S, Whitlock RP, Healey JS; on behalf of the LAAOS III Investigators. Heart failure after left atrial appendage occlusion: Insights from the LAAOS III randomized trial. Eur J Heart Fail. 2025 Feb;27(2):285-292. doi: 10.1002/ejhf.3536. Epub 2024 Nov 25. PMID 39586754
- [Derived] Whitlock RP, Belley-Cote EP, Paparella D, Healey JS, Brady K, Sharma M, Reents W, Budera P, Baddour AJ, Fila P, Devereaux PJ, Bogachev-Prokophiev A, Boening A, Teoh KHT, Tagarakis GI, Slaughter MS, Royse AG, McGuinness S, Alings M, Punjabi PP, Mazer CD, Folkeringa RJ, Colli A, Avezum A, Nakamya J, Balasubramanian K, Vincent J, Voisine P, Lamy A, Yusuf S, Connolly SJ; LAAOS III Investigators. Left Atrial Appendage Occlusion during Cardiac Surgery to Prevent Stroke. N Engl J Med. 2021 Jun 3;384(22):2081-2091. doi: 10.1056/NEJMoa2101897. Epub 2021 May 15. PMID 33999547